CLINICAL TRIAL: NCT00257218
Title: A Study on Effect of Health Promotion for Prevention NIDDM in People With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 9461701008
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2005-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Behavioral: Life style modification

SUMMARY:
OBJECTIVE - The role of health promotion for patients with impaired fasting glucose on preventing or delay the progression of diabetes mellitus has not been widely investigated in Taiwan. The purposes of this study are to explore the nature history of prediabetes, to evaluate the incidence of DM in prediabetes and to establish the cohort of people with prediabetes. Further study will be based on this cohort to evaluate the effect of health promotion and to compare the concentration of certain protein in their serum, such as adiponectin.

RESEARCH DESIGN AND METHODS -A total of 600 subjects aged 40-60 years with impaired fasting glucose (100-125 mg/dl) were randomly selected from the Peng-Hu clinics during January 2003 and December 2003. Anthropometric, biochemical, and metabolic characteristics will be measured, including weight, height, waist circumference, oral glucose tolerance test, triglyceride, high and low density cholesterol, blood pressure and insulin resistance etc. A questionnaire interviews with subjects regarding demographic characteristics is also performed. 300 subjects will receive education of health promotion. Simultaneously, 150 subjects with normal fasting plasma glucose (<100 mg/dl) will selected for comparison.

Statistical Analysis - Descriptive data will be described as means and SDs for continuous variables, and analysis of variance (ANOVA) and Chi-square tests were used for assessing the significances. Bonferroni method was used for post-hoc comparison in ANOVA. Multiple linear regressions were used for predicting determinants of FPG. We tested the variables scales in this study for multicollinearity by correlation matrix and VIF (variance inflation factor). Odds ratios (ORs) and the 95% confidence interval (CI) were calculated to estimate the relative risk of diabetes mellitus by logistic regression model. A p-value below 0.05 was considered significant. The statistical analyses were performed with SPSS statistical Package.

ELIGIBILITY:
Inclusion Criteria:

* fasting glucose level 100-125mg/dl
* OGTT 2hr glucose level 140-199 mg/dl

Exclusion Criteria:

* established diabetes mellitus: use of diabetic medication, fasting glucose >=126 mg/dl, OGTT 2ht glucose level >=200mg/dl

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000
Dates: Start 2006-01

PRIMARY OUTCOMES:
Incidence of diabetes mellitus

SECONDARY OUTCOMES:
insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Nan Wei, Ph.D., Principal Investigator — Chia Nan University of Pharmacy and Science
Locations (1):
- Chia Nan University of Pharmacy and Science, Tainan, Taiwan